CLINICAL TRIAL: NCT06026644
Title: Health-Related Quality of Life Outcomes in Patients With Aggressive B-Cell Lymphomas Treated With CAR-T Cell Therapy in Real Life: A Multicenter Prospective Observational Study
Brief Title: Health-Related Quality of Life Outcomes in Patients With Aggressive B-Cell Lymphomas Treated With CAR-T Cell Therapy in Real Life
Acronym: LNH012
Status: Active, not recruiting | Type: Observational
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Other Study IDs: GIMEMA _QoL _CAR-T
Record Dates: First submitted 2023-07-05; First posted 2023-09-07 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2023-07

CONDITIONS: DLBCL - Diffuse Large B Cell Lymphoma
MeSH Terms: conditions — Dendritic Cell Sarcoma, Interdigitating

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Quality of life assessment: Quality of life questionnaires

SUMMARY:
This study will ultimately aim at providing the scientific community with patient-reported health status data that will contribute facilitate decision-makings. Short- and long-term HRQoL and symptoms will be evaluated in a longitudinal fashion over time to improve the understanding of the impact of the disease and CAR-T cell therapy on patients-wellbeing, symptom burden and daily functioning. This study will capture useful information on the impact of treatment toxicity, the burden of procedures on HRQoL outcomes. The planned collection of PRO and physician-reported adverse events ad early time point will help to compare and integrate these two points of view in healthcare assessment.

DETAILED DESCRIPTION:
Quality of life assessment

ELIGIBILITY:
Inclusion Criteria:

* Patients with diffuse large B-cell lymphoma (DLBCL) not otherwise specified, primary mediastinal large B-cell lymphoma, high grade B-cell lymphoma, and DLBCL transformed by indolent lymphoma and mantle cell lymphoma.
* Scheduled to received CAR-T cell product.
* Having a baseline PRO assessment.
* Adult patients (≥ 18 years old).
* Written informed consent provided.

Exclusion Criteria:

* Having any documented or psychiatric or neurological disorder which may interfere with self-reported HRQoL assessment.
* Not able to read and understand local language.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Aggressive B-Cell Lymphomas Treated with CAR-T Cell Therapy
Sampling Method: Non-Probability Sample
Enrollment: 170 (Estimated)
Dates: Start 2022-06-29 (Actual); Primary Completion 2024-02-15 (Actual); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
The proportion of patients with a clinically meaningful improvement in the fatigue score of the PROMIS- Fatigue questionnaire | at 12 months
  To assess the proportion of patients with a clinically meaningful improvement in the fatigue score of the PROMIS- Fatigue questionnaire

SECONDARY OUTCOMES:
The proportion of patients with a clinically meaningful improvement in the scales of the EORTC QLQ-C30 questionnaire | at 12 months
  To assess the proportion of patients with a clinically meaningful improvement in the scales of the EORTC QLQ-C30 questionnaire
The time to improvement in the PROMIS-Fatigue score | After 2 years from date of registration
  To assess the time to improvement in the PROMIS-Fatigue score
The time to improvement in the EORTC QLQ-C30 questionnaires | After 2 years from date of registration
  To assess the time to improvement in the EORTC QLQ-C30 questionnaires
The time to improvement in the QLQ-NHL-HG29 questionnaires | After 2 years from date of registration
  To assess the time to improvement in the QLQ-NHL-HG29 questionnaires
The trajectories over time (up to 24 months) of the mean scores from the PROMIS-Fatigue questionnaire. | After 2 years from date of registration
  To estimate the trajectories over time (up to 24 months) of the mean scores from the PROMIS-Fatigue questionnaire.
The trajectories over time (up to 24 months) of the mean scores from the EORTC QLQ-C30 questionnaire. | After 2 years from date of registration
  To estimate the trajectories over time (up to 24 months) of the mean scores from the EORTC QLQ-C30 questionnaire.
The trajectories over time (up to 24 months) of the mean scores from the EORTC QLQ-NHL-HG29 questionnaire. | After 2 years from date of registration
  To estimate the trajectories over time (up to 24 months) of the mean scores from the EORTC QLQ-NHL-HG29 questionnaire.
Short-term (ie., day+10) patient-reported symptomatic toxicities by a core set of items from the PRO-CTCAE Item Library, and comparing them with those reported by the treating physicians. | After + 10 day for infusion
  To assess short-term (ie., day+10) patient-reported symptomatic toxicities by a core set of items from the PRO-CTCAE Item Library, and comparing them with those reported by the treating physicians
The impact of CAR-T cell therapy on cognitive impairment as measured by the PROMIS Cognitive Function short form 8a questionnaire. | After 2 years from date of registration
  To investigate the impact of CAR-T cell therapy on cognitive impairment as measured by the PROMIS Cognitive Function short form 8a questionnaire.
The long-term HRQoL and fatigue profile of patients with that of their peers from the general population, using the PROMIS-Fatigue questionnaire. | After 12 and 24 months from date of registration
  To compare the long-term HRQoL and fatigue profile of patients with that of their peers from the general population, using the PROMIS-Fatigue questionnaire.
The long-term HRQoL and fatigue profile of patients with that of their peers from the general population, using the EORTC QLQ-C30 questionnaire. | After 12 and 24 months from date of registration
  To compare the long-term HRQoL and fatigue profile of patients with that of their peers from the general population, using the EORTC QLQ-C30 questionnaire.
Factors predicting response to therapy and survival outcomes | After 2 years from date of registration
  To identify pretreatment factors predicting response to therapy and survival outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Alice Di Rocco, Principal Investigator — Aou Policlinico Umberto I - Dipartimento Di Medicina Traslazionale - Sezione Ematologia
Locations (13):
- Italy (13):
  - Aou Di Bologna - Policlinico S. Orsola-malpighi - Uoc Ematologia, Bologna
  - Asst Degli Spedali Civili Di Brescia - Ssvd Centro Trapianti Midollo Per Adulti - Cattedra Di Ematologia, Brescia
  - AOU Careggi - SOD terapie cellulari e Medicina Trasfusionale, Florence
  - Irccs Aou San Martino - Genova - Uo Ematologia E Trapianti, Genova
  - Fondazione Irccs "Istituto Nazionale Tumori" - Milano - Sc Ematologia, Milan
  - Ao Ospedali Riuniti Villa Sofia Cervello - Palermo - Uo Ematologia Ad Indirizzo Oncologico, Palermo
  - Asl Pescara, Presidio Ospedaliero 'Spirito Santo' - Uoc Ematologia Clinica, Pescara
  - Aou Pisana - Uo Ematologia Universitaria, Pisa
  - Aou Policlinico Umberto I - Dipartimento Di Medicina Traslazionale - Sezione Ematologia, Roma
  - Ististuto Clinico Humanitas - Rozzano - Uo Oncologia Medica Ed Ematologia, Rozzano
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia - Università Degli Studi Di Torino, Torino
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia 2, Torino
  - Aulss 8 Berica - Ospedale Di Vicenza - Uoc Ematologia, Vicenza